CLINICAL TRIAL: NCT06976242
Title: Comparison Of The Effectiveness Of Elastic Resistance Versus Free Weight Training Of Gluteus Medius In Improving Pain, Strength, And Overall Gait Speed In Patients With Chronic Non-Specific Low Back Pain: Randomized Controlled Trial
Brief Title: Comparison Of The Effectiveness Of Elastic Resistance Versus Free Weight Training Of Gluteus Medius In Improving Pain, Strength, And Overall Gait Speed In Patients With Chronic Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/001
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain
Keywords: Gluteus Medius; Low Back Pain; Chronic Non-Specific Low Back Pain; Exercise Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an elastic resistance training group or a free weight training group to compare outcomes related to pain, strength, and gait speed.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and assessors performing pre- and post-intervention evaluations will be blinded to group allocation to reduce bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic Resistance Training with Conventional Training (Experimental): The participants in this group will receive elastic resistance training with conventional training. The intervention would be given 5 times per week on alternate days for 4 weeks. Each exercise session will be given in 2sets of 8 repetitions each set.
  Interventions: Procedure: Elastic Resistance Training; Procedure: Conventional Training
- Free Weight Training along with Conventional Training (Active Comparator): The participants in this group will receive free weight training along with conventional training. The intervention frequency will be the same as group A (5 times/week for 4 weeks). Each exercise session will be given in 2 sets of 8 repetitions each set.
  Interventions: Procedure: Free Weight Exercises; Procedure: Conventional Training

INTERVENTIONS:
Procedure: Elastic Resistance Training — The type of resistance exercises in which the participants use the Thera Band of yellow and red colours (weight about 2-2.5 kg with full elongation) for resistance training
  Other Names: Resistance Band Training, Theraband Exercise
  Arms: Elastic Resistance Training with Conventional Training
Procedure: Free Weight Exercises — The type of resistance exercises in which the participants use weight cuffs (weight 2-2.5 kg) tied to their lower leg for resistance training
  Arms: Free Weight Training along with Conventional Training
Procedure: Conventional Training — The conventional training includes side-lying hip abductions, standing weighted abductions, and lateral step-ups exercises.

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of elastic resistance training and free weight training in strengthening the gluteus medius muscle among patients with chronic non-specific low back pain. Weakness in the gluteus medius can contribute to pelvic instability and altered gait patterns, which may exacerbate low back pain. While both elastic resistance and free weight exercises are commonly used in rehabilitation, there is limited evidence comparing their relative benefits in this population. This study evaluates improvements in pain, muscle strength, and overall gait speed following each intervention. The findings will help guide clinicians in choosing the most effective and accessible strengthening method for patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
The gluteus medius plays a vital role in pelvic stabilization and maintaining proper gait mechanics. Dysfunction or weakness in this muscle is frequently associated with chronic non-specific low back pain, a condition affecting a significant proportion of the population. Rehabilitation strategies that target the gluteus medius are crucial for restoring lumbar-pelvic stability, optimizing functional movement, and reducing pain.

Free weight training, using equipment like dumbbells and barbells, is a traditional method to enhance muscle strength and improve neuromuscular coordination. However, it often requires proper supervision to avoid injury due to the need for controlled movements and joint stability. On the other hand, elastic resistance training, which employs tools like resistance bands or tubes, offers a safer, cost-effective, and portable alternative. It allows progressive resistance throughout the range of motion, matching the user's strength curve and facilitating home-based exercise programs.

This randomized controlled trial is designed to compare these two training modalities, which are elastic resistance versus free weights in terms of their effectiveness at improving gluteus medius strength, reducing low back pain, and enhancing gait speed in patients with chronic non-specific low back pain. The trial includes baseline and post-intervention assessments using validated clinical tools for measuring pain, strength, and gait speed.

The goal is to determine which intervention yields greater clinical benefit and offers a more practical approach for implementation in therapeutic settings, especially for populations with limited access to conventional gym equipment. The findings could contribute valuable evidence to inform clinical decision-making in physical therapy and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-60 years
2. Both males and females of any race and ethnicity
3. Musculoskeletal condition that affects the gluteus Medius of hip
4. MMT for gluteus medius is 3 or less than 3
5. chronic stage of nonspecific low back pain
6. Cognitively intact (mini mental scale) and able to walk 10 meters with or without support.
7. Volunteer participations.

Exclusion Criteria:

1. Post-surgical conditions like TKR, THR.
2. Any contraindication to exercise.
3. Female individuals who have muscular weakness due to pregnancy
4. Any neurological conditions (myopathies, neuropathies) causing muscular weakness
5. Chronic low back pain in which Gluteus Medius weakness is not measurable.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity | Baseline and at 4 weeks post-intervention
  Pain will be assessed using the Numeric Pain Rating Scale (NPRS), a self-reported 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain).
Change in Gluteus Medius Muscle Strength | Baseline and at 4 weeks post-intervention
  Muscle strength will be measured using a manual muscle testing to assess isometric strength of the gluteus medius. A system of manually testing weakness of muscles by assuming different positions and performing movements against gravity or gravity eliminated depending on the strength of the and 5 indicates the muscle can hold anti-gravity position against maximum resistance.
Change in Overall Gait Speed | Baseline and at 4 weeks post-intervention
  Gait speed will be measured using the 10-Meter Walk Test (10MWT), recorded in meters per second (m/s).

CONTACTS AND LOCATIONS:
Overall Officials: Gulab Noor, MSPT, Principal Investigator — Institute of Physical Medicine and Rehabilitation, Khyber Medical University Peshawar; Dr Hazrat Bilal, PhD*, Principal Investigator — Institute of Physical Medicine and Rehabilitation, Khyber Medical University Peshawar
Locations (1):
- Rehman Medical Institute, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interested in the stated study area after its proper monitoring. Data or samples shared will be coded, with no PHI included. Prior permission of the investigators, participants and concerned departments will be obtained.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 12 months after article publication.
Access Criteria: Access can be requested by qualified researchers through proper approval of the investigators.

REFERENCES:
- [Background] Roelker SA, Kautz SA, Neptune RR. Muscle contributions to mediolateral and anteroposterior foot placement during walking. J Biomech. 2019 Oct 11;95:109310. doi: 10.1016/j.jbiomech.2019.08.004. Epub 2019 Aug 9. PMID 31451199
- [Background] Ventura JD, Klute GK, Neptune RR. Individual muscle contributions to circular turning mechanics. J Biomech. 2015 Apr 13;48(6):1067-74. doi: 10.1016/j.jbiomech.2015.01.026. Epub 2015 Feb 2. PMID 25700608
- [Background] Kasitinon D, Li WX, Wang EXS, Fredericson M. Physical Examination and Patellofemoral Pain Syndrome: an Updated Review. Curr Rev Musculoskelet Med. 2021 Dec;14(6):406-412. doi: 10.1007/s12178-021-09730-7. Epub 2021 Oct 29. PMID 34713383
- [Background] Bauer CM, Rast FM, Ernst MJ, Meichtry A, Kool J, Rissanen SM, Suni JH, Kankaanpaa M. The effect of muscle fatigue and low back pain on lumbar movement variability and complexity. J Electromyogr Kinesiol. 2017 Apr;33:94-102. doi: 10.1016/j.jelekin.2017.02.003. Epub 2017 Feb 13. PMID 28226298
- [Background] Lanza MB, Rock K, Marchese V, Addison O, Gray VL. Hip Abductor and Adductor Rate of Torque Development and Muscle Activation, but Not Muscle Size, Are Associated With Functional Performance. Front Physiol. 2021 Oct 14;12:744153. doi: 10.3389/fphys.2021.744153. eCollection 2021. PMID 34721067
- [Background] Sheahan PJ, Diesbourg TL, Fischer SL. The effect of rest break schedule on acute low back pain development in pain and non-pain developers during seated work. Appl Ergon. 2016 Mar;53 Pt A:64-70. doi: 10.1016/j.apergo.2015.08.013. Epub 2015 Sep 10. PMID 26674405
- [Background] Khayambashi K, Ghoddosi N, Straub RK, Powers CM. Hip Muscle Strength Predicts Noncontact Anterior Cruciate Ligament Injury in Male and Female Athletes: A Prospective Study. Am J Sports Med. 2016 Feb;44(2):355-61. doi: 10.1177/0363546515616237. Epub 2015 Dec 8. PMID 26646514
- [Background] Butowicz CM, Ebaugh DD, Noehren B, Silfies SP. VALIDATION OF TWO CLINICAL MEASURES OF CORE STABILITY. Int J Sports Phys Ther. 2016 Feb;11(1):15-23. PMID 26900496
- [Background] Qiu J, Zhou T, Jin H, Pan Y, Qian T, Xue C, Xia W, Shi H, An B. Effect of adding hip exercises to general rehabilitation treatment of knee osteoarthritis on patients' physical functions: a randomized clinical trial. BMC Sports Sci Med Rehabil. 2023 Nov 23;15(1):158. doi: 10.1186/s13102-023-00772-7. PMID 37996958
- [Background] Lorenzetti S, Ostermann M, Zeidler F, Zimmer P, Jentsch L, List R, Taylor WR, Schellenberg F. How to squat? Effects of various stance widths, foot placement angles and level of experience on knee, hip and trunk motion and loading. BMC Sports Sci Med Rehabil. 2018 Jul 17;10:14. doi: 10.1186/s13102-018-0103-7. eCollection 2018. PMID 30026952
- [Background] Psilander N, Eftestol E, Cumming KT, Juvkam I, Ekblom MM, Sunding K, Wernbom M, Holmberg HC, Ekblom B, Bruusgaard JC, Raastad T, Gundersen K. Effects of training, detraining, and retraining on strength, hypertrophy, and myonuclear number in human skeletal muscle. J Appl Physiol (1985). 2019 Jun 1;126(6):1636-1645. doi: 10.1152/japplphysiol.00917.2018. Epub 2019 Apr 11. PMID 30991013